CLINICAL TRIAL: NCT02256566
Title: Cognitive Training for Mood and Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 14-0994
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Major Depressive Disorder; Depression; Bipolar Disorder; Post-traumatic Stress Disorder; Generalized Anxiety Disorder; Social Phobia
Keywords: cognitive training; depression; bipolar depression; anxiety; ptsd; generalized anxiety; social phobia
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Bipolar Disorder; Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Phobia, Social; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- emotional memory training exercise (Experimental): study training exercise - Emotional Faces Memory Task (EFMT)
  Interventions: Behavioral: emotional memory training exercise
- memory training exercise (Active Comparator): an active control exercise (CT)
  Interventions: Behavioral: memory training exercise

INTERVENTIONS:
Behavioral: emotional memory training exercise
  Arms: emotional memory training exercise
Behavioral: memory training exercise
  Arms: memory training exercise

SUMMARY:
The purpose of this study is to investigate the effects of a computerized cognitive training program (an attention and memory exercise performed on a computer) on thinking and memory in individuals with mood and anxiety disorders, and to begin to test whether this training affects symptoms of depression or anxiety.

DETAILED DESCRIPTION:
The objective of this research protocol is to collect feasibility and pilot data investigating the efficacy of a computerized cognitive training paradigm. The training paradigm aims to enhance cognitive control for emotional information-processing and reduce the negative affective biases observed among those experiencing mood and anxiety symptoms and disorders. This protocol will also investigate whether improvements in cognitive control and affective bias are associated with changes in mood and anxiety symptoms. Participants will undergo 6 weeks of cognitive training sessions, with three sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* Primary, current Axis I diagnosis of a mood disorder (e.g., major depressive disorder (MDD); bipolar disorder, currently depressed) or anxiety disorder (PTSD; Generalized Anxiety Disorder (GAD); Social Phobia) according to DSM-IV criteria and SCID-IV diagnosis OR must be free of any psychiatric condition (for the healthy volunteer group)
* Age 18-80
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process

Exclusion Criteria:

* A history of drug or alcohol abuse or dependence (DSM-IV criteria) within the previous 6 months
* Visual impairment that would affect the ability to observe the computerized exercises
* Motor impairment that would affect the ability to provide a response by quickly pressing a button
* Patients with mood congruent or mood incongruent psychotic features
* Primary, current Axis I diagnosis other than MDD, Bipolar Disorder (currently depressed), PTSD, GAD or Social Phobia
* The presence of axis II personality disorder psychopathology that, in the opinion of the investigator, will interfere with study participation
* Acute suicidal or homicidal risk (evidenced by suicidal or homicidal attempt within 6 months of screening)
* Pregnancy in women. Pregnant women are excluded from the study because research has shown that hormonal changes that occur during pregnancy can mimic and/or influence symptoms of depression. Including patterns of mood and cognition. These mood and cognitive changes could mask the effect of the cognitive training in this study, so pregnant women will be excluded for that reason. A urine pregnancy test will be administered at screening
* Enrolled participants can be currently taking standard antidepressant or mood stabilizer medication regimens, or benzodiazepine treatment for sleep as needed but not exceeding 3 nights per week. Medication regimens must be stable at the time of study enrollment (i.e., no medication has been started within 8 weeks, stopped within 6 weeks or titrated up or down within 4 weeks of study entry). No medications will be started or discontinued for the purpose of enrollment into the study
* Subjects must exhibit no or only moderate alcohol use during study participation. Subjects with current excessive use of alcohol (> 8 ounces/day) or participants abusing substances will be ineligible for participation, as such drug use could confound the results. A urine toxicology test will be administered at screening to test for drugs of abuse
* Participants exhibiting depression symptoms in the severe range (Ham-D > 27) will be excluded from participation as an investigational study such as this may not be suitable
* Participants exhibiting chronic MDD episodes (defined as a current episode lasting 5+ years) will be excluded from participation as an investigational study such as this may not be suitable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
Proportion of completers to measure feasibility | week 6
  comparing the proportion of completers (15-18 sessions) between the in-person participants and the participants completing the exercise on their own computers

SECONDARY OUTCOMES:
Change in Depression Symptom Severity | baseline and week 6
  Depression symptom severity comparison at week 6 to baseline as measured by the Hamilton Depression Rating Scale (Ham-D) and Quick Inventory of Depressive Symptoms (QIDS-C)
Change in Anxiety Symptom Severity | baseline and week 6
  Anxiety symptom severity comparison at week 6 to baseline as measured by the Hamilton Anxiety Rating Scale (Ham-A) and Treatment Outcome PTSD Scale (TOP-8)
Change in Negative Affective Bias | baseline and week 6
  Negative affective bias comparison at week 6 to baseline as measured by the Self-referential Information Processing Task, Affective Go/No-Go, Emotional Stroop, Emotion Faces Recognition Task, Cognitive Style Questionnaire, Ruminative Responses Scale, and Attention Bias Variability Task
Change in Neurocognition | baseline and week 6
  neurocognition comparison at week 6 to baseline using Digit Span, Letter-Number Sequencing, Hopkins Verbal Learning Test, and Intra-Extra Dimensional Set-Shifting

CONTACTS AND LOCATIONS:
Overall Officials: Brian Iacoviello, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States